CLINICAL TRIAL: NCT04742920
Title: The Onyx™ Trial For The Embolization Of The Middle Meningeal Artery For Chronic Subdural Hematoma (OTEMACS)
Brief Title: The Onyx™ Trial For The Embolization Of The Middle Meningeal Artery For Chronic Subdural Hematoma
Acronym: OTEMACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The DSMB recommended to stop the study after the interim analysis, as the results shown a superiority of the embolization arm. 247 patient were finally enrolled.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL20_0362
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hematoma, Subdural, Chronic; Brain Diseases; Central Nervous System Diseases; Wounds and Injuries
Keywords: Chronic Subdural Hematoma; Middle Meningeal Artery; Embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Brain Diseases; Central Nervous System Diseases; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMA embolization group (Other): MMA embolization procedure with Onyx™ in addition to standard (surgical/conservative) management
  Interventions: Device: Middle Meningeal Artery Embolization
- Control group (Other): Standard (surgical/conservative) Management alone
  Interventions: Procedure: Standard Management

INTERVENTIONS:
Device: Middle Meningeal Artery Embolization — MMA embolization using the Onyx™ non-adhesive liquid embolic agent within 72 hours after randomization in addition to standard management
  Arms: MMA embolization group
Procedure: Standard Management — Procedure : Surgical Management Surgical evacuation of the subdural hematoma
  Other: Conservative Management Standard medical management: drug treatment and/or observation
  Arms: Control group

SUMMARY:
Middle meningeal artery (MMA) embolization via a minimally invasive endovascular approach might increase the likelihood of resolution and might prevent reaccumulation of Chronic Subdural Hematoma (CSDH). The purpose of the OTEMACS Trial is to assess the safety and effect on recurrence rate and functional outcome of endovascular treatment in patients with CSDH.

DETAILED DESCRIPTION:
The OTEMACS study is a prospective, multicenter clinical trial with randomized treatment allocation, open label treatment and blinded endpoint evaluation (PROBE), designed to demonstrate that MMA embolization via a minimally invasive endovascular approach combined with standard (surgical/conservative) management is superior to standard management alone, in reducing the rate of CSDH-related surgical interventions and the recurrence rate in patient with CSDH at 90 days.

Eligible symptomatic CSDH patients will be randomly assigned, in a 1:1 ratio, to receive either surgical treatment plus an adjuvant MMA embolization (ST+MMAE group; the Experimental arm) or surgical treatment alone (ST group; the Control arm).

Eligible symptomatic nonsurgically treated patients with CSDH will be randomized, in a 1:1 ratio, to MMA embolization (MMAE group; the Experimental arm) or conservative management (CM group; the Control arm).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at inclusion (no upper age limit).
* CSDH confirmed on cranial imaging (e.g. CT/magnetic resonance imaging [MRI]), as documented by a radiologist.
* One or more symptoms attributable to CSDH including headache, cognitive impairment, gait instability, seizure, mild focal neurologic deficit, speech disturbance, or decreased consciousness.
* No significant pre-morbid disability (baseline mRS score ≤3).
* Decision of conventional therapy (neurosurgeon blinded to the randomization group)
* Patient or patient's representative has received information about the study and has signed and dated the appropriate Informed Consent Form, or fulfilling the criteria for emergency consent.

Exclusion Criteria:

* CSDH developing with underlying conditions: vascular lesions, brain tumor, arachnoid cyst, or spontaneous intracranial hypotension.
* CSDH that have a focal location (confined to the frontal or temporal base or the interhemispheric space without cerebral convexity involvement), is 10 mm or less in thickness, or have no mass effect (cortical flattening or midline shifting).
* Known absence of vascular access or any local cause prohibiting femoral catheterization.
* Known contrast or endovascular or anesthetic product allergy or contraindications.
* Any contraindications to the use of the Onyx™.
* Female who is known to be pregnant or lactating at time of admission.
* Patient presenting severe or fatal co-morbidities or Life expectancy under 6 months that will likely interfere with improvement or follow-up or that will render the procedure unlikely to benefit the patient.
* Patient unable to be present or available for follow-up
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations (e.g. severe dementia).
* Current participation in another investigational drug or device study.
* Major patients under court protection, guardianship or curatorship.
* Not be affiliated to a French social security system or a beneficiary of such a system

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Recurrence rate in the Experimental group vs. the Control group | Within 90 days
  The recurrence of CSDH is defined by:
  * radiological remaining of the hematoma with thickness > 10 mm in the ipsilateral subdural space with or without any clinical presentation at 90 days (+/- 14 days) after the randomization OR
  * revision surgery (in surgical group) / surgical rescue (non-surgical group) for hematoma reaccumulation (as assessed

SECONDARY OUTCOMES:
Mortality rates at discharge | Within 7 days
Major disabling stroke at discharge | Within 7 days
Incidence of procedure-related and device-related serious adverse events (PRSAEs and DRSAEs) | Through 24 hours (-6/+24 hours) post endovascular treatment
Rate of recurrence of CSDH requiring revision surgery (in surgical group) or surgical rescue (in non-surgical group) | Within 90 days
Change in hematoma volume (HV) in the Experimental group vs. the Control group | At 90 days
Shift on the modified Rankin Scale (mRS) score in the Experimental group vs. the Control group | At 90 days
Proportion of patients with good functional outcome, defined as mRS 0-2 | At 90 days
Proportion of patients with favorable functional outcome, defined as mRS 0-3 | At 90 days
Degree of disability (shift on the mRS combining scores of 5 and 6) | At 90 days
Distribution of utility weighted mRS (UW mRS) | At 90 days
Quality of life assessed by the EuroQol (Quality of life) EQ-5D scale | At 90 days
Quality of life assessed by the Barthel Index | At 90 days
Length of hospital stay for neurosurgery. | within 90 days
Incidence of all-cause mortality | At 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COSTALAT, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (6):
- France (6):
  - CHU de Bordeaux Hôpital Pellegrin, Bordeaux
  - CHU Lyon, Bron
  - CHU de Dijon, Dijon
  - Chu de Montpellier - Gui de Chauliac, Montpellier
  - CHU de Nîmes, Nîmes
  - CHU de Toulouse Hôpital Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No